CLINICAL TRIAL: NCT00002209
Title: Multiple Ascending Dose Pharmacokinetics of CPI-1189 (LU 02-584) in Fasted, HIV Infected, Male Volunteers on Combined Reverse Transcriptase and Protease Inhibitor Therapy
Brief Title: Safety and Effectiveness of CPI-1189 in HIV-Infected Males on Combination Anti-HIV Drug Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centaur Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 289A; CPI001189-MAD01
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-12

CONDITIONS: AIDS Dementia Complex; HIV Infections
Keywords: Dose-Response Relationship, Drug; Drug Therapy, Combination; AIDS Dementia Complex; Zidovudine; Lamivudine; Indinavir; Reverse Transcriptase Inhibitors
MeSH Terms: conditions — AIDS Dementia Complex; HIV Infections | interventions — CPI 1189

INTERVENTIONS:
Drug: CPI-1189

SUMMARY:
The purpose of this study is to see if it is safe to give multiple doses of CPI-1189 to HIV-infected, otherwise healthy, males. The study will also look at how CPI-1189 affects the levels of HIV, T cells (cells in the body that help fight infection), and three anti-HIV drugs (zidovudine, lamivudine, and indinavir) in the blood.

Advanced HIV infection can cause AIDS dementia (brain damage due to HIV leading to losses of memory and muscle control). CPI-1189 may be able to postpone AIDS dementia or slow it down.

DETAILED DESCRIPTION:
Late-stage HIV infection can cause AIDS dementia (brain damage due to HIV leading to losses of memory and muscle control). CPI-1189 may be able to postpone AIDS dementia or slow it down.

In this randomized, double-blind study, 48 HIV-infected, otherwise healthy, male volunteers receive either multiple-dose CPI-1189 or placebo by mouth for 15 consecutive days. Each dosing group begins 6 weeks following the start of the preceding group. Volunteers enter the study site the night before dosing on Days 1 and 15 and remain at the study site for 72 hours following dosing. Throughout the study, volunteers have physical exams and donate samples of blood, urine, cerebrospinal fluid, and sperm.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are an HIV-positive man who is otherwise in good health.
* Are 18-50 years old.
* Have a CD4 count of 75-500 cells/mm3.
* Are currently taking zidovudine (ZDV), lamivudine (3TC), and indinavir (IDV).

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48

CONTACTS AND LOCATIONS:
Locations (1):
- MDS Harris, Phoenix, Arizona, United States